CLINICAL TRIAL: NCT02231255
Title: Switch Post Marketing Surveillance Study in Patients With Idiopathic Parkinson's Disease
Brief Title: Post Marketing Surveillance Study in Patients With Idiopathic Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 248.517
Record Dates: First submitted 2014-09-02; First posted 2014-09-04 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Pramipexole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Idiopathic Parkinson's disease patients
  Interventions: Drug: Sifrol®

INTERVENTIONS:
Drug: Sifrol®

SUMMARY:
Documentation of the effect of an direct or overlapping switch from another dopamine agonist to Sifrol® on motor function, psychopathological disturbances and mood, assessment of the reasons for the switch and the reasons for using Sifrol®, equivalent doses at the end of the switch and tolerability of Sifrol® in ambulatory patients suffering from idiopathic Parkinson's disease under routine conditions

ELIGIBILITY:
Inclusion Criteria:

* Patients with Idiopathic Parkinson's disease who are planned to undergo a switch from another dopamine agonist to Sifrol®

Exclusion Criteria:

* Neurologists and psychiatrists are asked to consider the Summary of Product Characteristics (SPC) for Sifrol®

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Idiopathic Parkinson's disease patients recruited at office-based neurologists, psychiatrist or special neurology clinics
Sampling Method: Non-Probability Sample
Enrollment: 1216 (Actual)
Dates: Start 2002-02; Primary Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Reason for switch of therapy and reason for using Sifrol® | up to 8 weeks
  questionnaire
Type of switch (abrupt or overlapping) | up to 8 weeks
Changes in motor function by means of 5-points rating scale | up to 8 weeks
  Short Parkinson's Evaluation Scale (SPES)
Changes in psychopathological memory disturbances by means of 5- point rating scale | up to 8 weeks
  Short Parkinson's Evaluation Scale (SPES)
Changes in psychopathological thought disorder disturbances by means of 5- point rating scale | up to 8 weeks
  SPES score
Changes in psychopathological depression disturbances by means of 5- point rating scale | up to 8 weeks
  SPES score
Changes of mood on seven visual analogue scales (VASs) | up to 8 weeks
  assessed by patient
Equivalent doses of Sifrol® | after 8 weeks
  compared to previous treatment dosing, based on global clinical impression
Global assessment of efficacy by investigator on a 5-point rating scale | after 8 weeks

SECONDARY OUTCOMES:
Number of patients with adverse drug reactions | up to 8 weeks
Assessment of tolerability by investigator on a 5-point rating scale | after 8 weeks